CLINICAL TRIAL: NCT00535834
Title: Data Analysis for 00-C-0154, A Randomized Phase II Study of a PSA-based Vaccine in Patients With Localized Prostate Cancer Receiving Standard Radiotherapy
Brief Title: Studying Stored Samples From Patients With Localized Prostate Cancer Treated on Clinical Trial NCI-00-C-0154
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Other Study IDs: 999907214; 07-C-N214; CDR0000565972
Record Dates: First submitted 2007-09-25; First posted 2007-09-26 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage II prostate cancer; stage III prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Molecular Diagnostic Techniques

INTERVENTIONS:
Procedure: diagnostic procedure
Procedure: molecular diagnostic method
Procedure: protein expression analysis

SUMMARY:
RATIONALE: Studying samples of blood in the laboratory from patients before and after treatment may help doctors learn more about the effects of the treatment on cells.

PURPOSE: This clinical trial is studying samples collected from patients with localized prostate cancer who received treatment on clinical trial NCI-00-C-0154.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the formation of antibody complexes in serum samples taken before initiation of treatment and after completion of therapy in prostate cancer patients previously enrolled on clinical trial NCI-00-C-0154.
* Evaluate immunologic response.

Secondary

* Clone the underlying tumor antigens discovered through SEREX.

OUTLINE: Samples previously collected on clinical trial NCI-00-C-0154 (whole blood, serum, and peripheral mononuclear blood cells) are analyzed for immunologic responses and evidence of formation of anti-tumor antibodies. Western blot is used to detect any evidence of vaccine-induced autoantibody responses. If there is an indication of response, SEREX is used to clone the underlying antigens.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of localized adenocarcinoma of the prostate
* Received treatment on clinical trial NCI-00-C-0154

PATIENT CHARACTERISTICS:

* Consented the use of their collected blood cells for future research while enrolled on NCI-00-C-0154

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Immunologic response
Incidence of formation of antibody complexes in serum samples taken before initiation of treatment and after completion of therapy by western blot and SEREX

SECONDARY OUTCOMES:
Cloning of any underlying tumor antigens discovered in this process

CONTACTS AND LOCATIONS:
Overall Officials: James Gulley, MD, PhD, Principal Investigator — National Cancer Institute (NCI)